CLINICAL TRIAL: NCT04713852
Title: Predictive Value of SOFA and APACHE Scores for In-hospital Mortality in COVID-19 ICU Patients: a Longitudinal Single-center Study
Brief Title: Predictive Value of SOFA and APACHE Scores for In-hospital Mortality in COVID-19 ICU Patients
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Dr, Jessa Hospital
Other Study IDs: 2020-174
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the predictive value for in-hospital mortality of respectively the SOFA and Apache scores in a COVID-19 ICU cohort and to develop a new prediction model for COVID-19 patients admitted to the ICU from 13th of March 2020 until 17th of October 2020.

DETAILED DESCRIPTION:
The coronavirus disease (COVID-19), caused by the severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) emerged in December 2019 and has rapidly spread worldwide. The mortality of critical ill patients with COVID-19 has been reported variously as low as 11% and as high as 61%. The application of scoring systems can facilitate the effective evaluation by physicians to screen severe patients. At present, however, there are no specific scoring systems for the evaluation of COVID-19 patients. Scoring systems such as the Sequential Organ Failure Assessment (SOFA) score can help emergency or critical care physicians for prognosis and predicting mortality. The SOFA score described the condition of multiple organ dysfunction through several parameters, including oxygenation index, mean arterial pressure, Glasgow come scale, creatinine or urine volume, bilirubin, platelets for the respiratory, circulatory, neurological, renal, hepatogenic and coagulation systems respectively. The function of each organ system is scored from 0 to 4, and the individual SOFA scores are summed to a total score. Although SOFA was not initially designed to predict mortality, several studies reveal that SOFA could predict morbidity and mortality in severe ill patients.

Besides the SOFA score, the Acute Physiology and Chronic Health Evaluation (Apache II) scores was designed to measure the severity of disease of patients admitted to the ICU and to predict mortality. The Apache II score is calculated based on physiological measurements such as body temperature, mean arterial pressure, pH, heart and respiratory rate, Glasgow coma scale, oxygenation and blood parameters such as sodium, potassium, creatinine, hematocrit and white blood cell count. Recently, the Apache IV score is developed where additional parameters such as admission information, admission diagnosis and chronic health conditions were take into account.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients admitted to the ICU from 13th of March 2020 until 17th October 2020.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients admitted to the ICU from 13th of March 2020 until 17th October 2020.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Patients admitted from 13th march 2020 to 17th october 2020
  To predict the mortality based on the SOFA and Apache scores in critically ill ICU patients

SECONDARY OUTCOMES:
Predictive value | Patients admitted from 13th march 2020 to 17th october 2020
  Predictive value of DNR code, gender, BMI, hypertension, Diabetes, age, P/F ratio, anticoagulation and Rockwood Clinical Frailty index

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Belgium

REFERENCES:
- [Derived] Vandenbrande J, Verbrugge L, Bruckers L, Geebelen L, Geerts E, Callebaut I, Gruyters I, Heremans L, Dubois J, Stessel B. Validation of the Acute Physiology and Chronic Health Evaluation (APACHE) II and IV Score in COVID-19 Patients. Crit Care Res Pract. 2021 Jun 19;2021:5443083. doi: 10.1155/2021/5443083. eCollection 2021. PMID 34258059